CLINICAL TRIAL: NCT04315779
Title: Comparison of Conventional Laparoscopy and Natural Orifice Transluminal Endoscopic Surgery in the Surgical Treatment of Tubal Ectopic Pregnancy
Brief Title: Comparison of Two Different Approaches in the Surgical Treatment of Tubal Ectopic Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gokay Ozceltik, MD, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-2.1T/40
Record Dates: First submitted 2020-03-17; First posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Ectopic Pregnancy
Keywords: natural orifice transluminal endoscopic surgery; laparoscopy; ectopic pregnancy; minimally invasive surgery; quality of life; sexual function
MeSH Terms: conditions — Pregnancy, Ectopic | interventions — Salpingectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional laparoscopy (Active Comparator): In this arm, patients will be treated via conventional laparoscopy
  Interventions: Procedure: Salpingectomy
- Transvaginal natural orifice transluminal endoscopic surgery (Active Comparator): In this arm, patients will be treated via transvaginal natural orifice transluminal endoscopic surgery
  Interventions: Procedure: Salpingectomy

INTERVENTIONS:
Procedure: Salpingectomy — Patients will undergo removal of the affected tube

SUMMARY:
In this study we aim to compare conventional laparoscopy and natural orifice transluminal endoscopic surgery in the surgical treatment of ectopic pregnancy.

All the patients, with an indication of surgery for ectopic pregnancy, will be asked to participate in this clinical trial.

Indication of surgery will be based on clinical findings, ultrasound scans and serum hcg levels. There will be no exclusion criteria.

Duration of surgery, successful completion of the operation, intraoperative data and postoperative data will be collected.

All the patients will be asked to fill out quality of recovery-40 (QoR-40) questionnaire and 36-item short form health survey (SF-36) before surgery.

QoR-40 questionnaire will be repeated 24 hours after surgery and repeated every 24 hours until discharge. SF-36 will be repeated at 1-month follow-up visit. Patients will be also evaluated at postoperative 3-months, and female sexual function index will be asked to be filled-out.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age,
* Diagnosis of tubal ectopic pregnancy
* Patient's preference to undergo salpingectomy

Exclusion Criteria:

* Patients with contraindication to endoscopic surgery
* Refusal to sign informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-02-19 (Actual); Primary Completion 2021-02-19 (Estimated); Study Completion 2021-05-19 (Estimated)

PRIMARY OUTCOMES:
Successful completion of surgery as intended | Intraoperative, from the beginning to the end of surgical intervention
  The completion of the surgery with the route planned without having to change the surgical route
Operating time | Intraoperative
Reoperation rate | During follow-up, after surgery until hcg level drops below 5 U/L, up to 1 month
Complication rate | During follow-up, after surgery until hcg level drops below 5 U/L, up to 1 month

SECONDARY OUTCOMES:
Quality of Recovery-40 questionnaire | Preoperatively and Postoperative every 24 hours until discharge, expected to be up to 3 days following surgery
  The Quality of Recovery 40 questionnaire will be self-administered by patients at different time points
Quality of life change | Preoperative, Postoperative 1-month
  Short form 36 item health survery (SF-36) questionnaire will be self-administered by patients at different time points
Postoperative pain scores | Postoperative 2 hours, 6 hours, 12 hours, 24 hours, and every 24 hours until discharge (if the patient stays longer than 1 day at the hospital), , expected to be up to 3 days following surgery
  Postoperative pain will be assessed on a 10-cm visual analog scale at different time points
Sexual function | Postoperative 3 months
  Female sexual function index (FSFI) questionnaire will be self-administered by patients at postoperative 3-months
The need for additional analgesic use | Postoperative period until discharge, expected to be up to 3 days following surgery
  Patients will be routinely administered pethidine hydrochloride 3x50 mg parenteral on the day of surgery. Starting from postoperative day 1 patients will be administered paracetamol 500 mg oral upon their request. In case of inadequate pain relief and the need for additional analgesic use will ve recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University University Hospital, Department of Obstetrics and Gynecology, Bornova, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided